CLINICAL TRIAL: NCT07032350
Title: E-Tailored Pain Management Support for Dementia Family Caregivers
Brief Title: E-Tailored Pain Management Support for Dementia Family Caregivers: Feasibility of the PACE-app
Acronym: PACE-app
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Nai-Ching Chi, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202409203; AARGD-22-929062 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2025-06-19; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Care Giving Burden; Dementia; Chronic Pain; Pain Management; Palliative Care
Keywords: Dementia; Alzheimer Disease; Chronic Pain; Pain Management; Caregivers; Family Caregivers; Digital Health Intervention; eHealth; Web-based Intervention; Palliative Care; Home Care; Self-efficacy; Caregiver Stress; Caregiver Depression; Communication with Providers; Health Literacy; Rural Caregivers; Geriatrics; Aging; Cognitive Impairment; Pain Diary
MeSH Terms: conditions — Caregiver Burden; Dementia; Chronic Pain; Agnosia; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Active Comparator): Care recipients will continue receiving their regular pain care. Caregivers will complete outcome assessments only.
  Introductory Meeting (Baseline):
  Caregivers will attend a 1.5-hour meeting to complete informed consent and baseline REDCap surveys.
  Follow-up (Month 1 and Month 2):
  At 1-month and 2-month follow-ups, caregivers will independently complete REDCap surveys (~45 minutes per follow-up).
  Interventions: Behavioral: Usual Pain Management Care
- App Use Group (Experimental): Care recipients will continue receiving their regular pain care. Caregivers will use the PACE-app and complete outcome assessments.
  Introductory Meeting (Baseline):
  Caregivers will attend a 1.5-hour meeting to complete informed consent and baseline REDCap surveys.
  Intervention Period (Month 1):
  Caregivers will use the PACE-app for 1 month, complete a daily pain diary (5-10 minutes/day), and access weekly summary reports to share with providers.
  Post-Intervention (Month 1):
  Caregivers will complete REDCap surveys and participate in a 1.5-hour interview on their experience with the app (audio-recorded unless declined).
  Follow-up (Month 2):
  Caregivers will complete the same REDCap questionnaires to assess longer-term outcomes.
  Interventions: Other: Web-based pain management support tool

INTERVENTIONS:
Other: Web-based pain management support tool — The Pain Control Enhancement App (PACE-app) is a web-based tool designed to help family caregivers manage pain in persons with dementia. The app provides a brief screening to identify caregiver challenges and delivers tailored strategies, communication prompts for providers, and an educational resource library. It includes a digital pain diary for tracking daily pain, treatments, and urgent care use, with weekly reports that can be shared with healthcare providers. The app is accessible on any internet-connected device and designed for caregivers with varying levels of digital literacy.
  Other Names: PACE-app
  Arms: App Use Group
Behavioral: Usual Pain Management Care — Caregivers receive no new intervention; they manage their care recipient's pain according to standard practices. No access to the PACE-app is given during the study period.
  Other Names: Usual Care
  Arms: Usual Care Group

SUMMARY:
The goal of this clinical trial is to test whether a web-based application called the Pain Control Enhancement App (PACE-app) can support family caregivers in managing pain for their care recipients with dementia. The main questions it aims to answer are:

Is it feasible and acceptable for family caregivers to use the PACE-app?

Does using the PACE-app improve caregiver self-efficacy in pain management, adherence to pain treatments, communication with care providers, well-being, and their care recipient's pain conditions?

Researchers will compare caregivers who use the PACE-app to those who continue with their usual care practices to see if the app leads to better outcomes for both caregivers and care recipients.

Participants will:

Be randomly assigned to either the PACE-app group or a usual-care control group

Complete online surveys at baseline, 1 month, and 2 months

If assigned to the PACE-app group:

Use the PACE-app for 1 month to receive tailored pain management strategies and tools, and record their care recipient's pain in a digital diary

Participate in an interview about their experience with the app

All participation activities can be done remotely or in person.

DETAILED DESCRIPTION:
This randomized controlled trial will assess the feasibility, usability, and preliminary efficacy of the Pain Control Enhancement App (PACE-app), a web-based intervention designed to support family caregivers of persons with dementia in managing pain. The trial will also explore mechanisms through which the PACE-app may affect caregiver and care recipient outcomes.

Uncontrolled pain is common in people with dementia and presents unique challenges for caregivers, particularly those with limited access to specialized healthcare services. Family caregivers often lack adequate knowledge, skills, and support to manage pain effectively, contributing to suboptimal outcomes for both caregivers and care recipients.

The PACE-app provides tailored, technology-based pain management support that includes:

Screening of caregiver-specific challenges in pain management;

Personalized pain management strategies based on the screening results;

Communication tools to facilitate interactions with healthcare providers;

A digital pain diary for tracking care recipients' pain experiences.

A total of 60 family caregivers of people with dementia and chronic pain will be randomized 1:1 to either the PACE-app intervention group or a usual-care control group. Participants in the intervention arm will use the app for 1 month and complete outcome assessments at baseline, 1 month (post-intervention), and 2 months (follow-up). Participants in the control arm will continue their usual caregiving practices and complete assessments on the same schedule.

Primary outcomes include feasibility (recruitment, retention, adherence to study protocol) and acceptability (measured by app usage analytics and qualitative interviews). Secondary outcomes include changes in caregiver self-efficacy in pain management, adherence to prescribed pain treatments, caregiver burden, stress, depression, and communication with healthcare providers. The study will also examine potential mediators (caregiver knowledge, communication) and moderators (caregiver characteristics, dementia severity, caregiving relationship) of intervention effects.

Additionally, the study will explore whether improvements in caregiver outcomes are associated with better outcomes for care recipients, such as reduced pain intensity and fewer urgent care visits related to pain.

Data collected will inform refinement of the PACE-app and guide the design of a future large-scale efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Be a primary caregiver - (a family member, relative, or friend) of a person with dementia (or cognitive impairment) and chronic pain (lasting >3 months)'
* Be responsible for managing the care recipient's pain and pain treatments (including interpreting verbal or non-verbal pain communication).
* Be age 18 - 100.
* Be able to read and speak English.
* Have regular access to an electronic device (tablet, laptop, or computer) with internet connectivity (for using the app and participating in data collection).
* Be accessible by phone or email to schedule meetings.
* Be willing to commit to the full study duration and protocol.

Exclusion Criteria:

* Currently participating in another research study that could interfere with this intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Caregiver Self-Efficacy in Pain Management | Change from baseline to 1 month and 2 months
  Measured using the pain managment subscale of the Chronic Pain Self-Efficacy Scale (CPSS). This 7-item scale on a 10-100 scale assesses confidence in skills such as medication management, and non-pharmacological techniques. Higher scores indicate greater self-efficacy

SECONDARY OUTCOMES:
Caregiver adherence to Pain Treatments | Baseline, 1 month, 2 moths
  Measured using the 12-itemthe modified Adherence to Refills and Medications Scale (ARMS). Each item uses a 4-point Likert scale (1, never to 4, all the time). Higher scores (ranging 12 to 48) indicate poorer adherence. Cut-off scores define different adherence levels (e.g., <16=adherent, ≥20=non-adherent).
Caregiver Burden | Baseline, 1 month, 2 months
  Measured using the 12-item Zarit Burden Interview (ZBI-12). Responses use a 5-point scale (0, never to 4, nearly always). Higher scores (ranging 0 to 48) reflect greater burden.
Caregiver Stress | Baseline, 1 month, 2 months
  Measured using the 14-item Perceived Stress Scale (PSS-14). PSS-14 asks family caregivers about their feelings and thoughts over the past month, using a 5-point Likert scale (0 = never to 4 = very often). Higher scores (ranging from 0 to 56) indicate greater perceived stress.
Caregiver Depression | Baseline, 1 month, 2 months
  Measured using the 20-item Center for Epidemiologic Studies Depression Scale (CES-D). Answers are given on a 4-point scale (0, rarely to 3, most of the time). Total scores range from 0 to 60, with higher scores indicating more severe depressive symptoms.
Caregiver Knowledge in Pain Management | Baseline, 1 month, 2 months
  Modified 17-item scale originally developed for nurses, adapted for caregivers. Each item is rated on a five-point Likert scale (1 = completely disagree to 5 = completely agree). Higher total scores (ranging from 17 to 85) indicate less knowledge in pain management.
Caregiver Communication with Providers | Baseline, 1 month, 2 months
  Measured using modified Perceived Involvement in Care Scale (M-PICS). It contains 21 statements scored on a 5-point Likert scale (1, strongly disagree to 5, strongly agree). Total possible scores range from 20 (least perceived involvement) to 100 (most perceived involvement). Higher scores indicate greater perceived involvement in care.

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Ching Chi, PhD, MS, MSN, BSN, Principal Investigator — University of Iowa
Locations (1):
- College of Nursing, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy, individual participant data (IPD) collected in this study will not be shared with other researchers. Only aggregated study results will be published.